CLINICAL TRIAL: NCT02732093
Title: Does Stellate Ganglion Block Decrease Stress Response of Intubation?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abdelraheem elawamy, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: irb00008718/654
Record Dates: First submitted 2016-04-05; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Intubation; Stellate Ganglion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stellate block (Active Comparator): patients in this arm will receive ultrasonographic guided left stellate block with 6 ml of lidocaine 2% after routine induction of general anesthesia and before endotracheal intubation
  Interventions: Procedure: stellate block; Drug: lidocaine 2%
- control (Placebo Comparator): patients in this arm will receive ultrasonographic guided left stellate block with 6 ml normal saline (Na.Cl 0.9%) (control group) after routine induction of general anesthesia and before endotracheal intubation
  Interventions: Procedure: stellate block; Drug: Na.Cl 0.9% (placebo)

INTERVENTIONS:
Procedure: stellate block
  Other Names: cervicothoracic ganglion block
Drug: Na.Cl 0.9% (placebo)
  Arms: control
Drug: lidocaine 2%
  Arms: stellate block

SUMMARY:
In this study investigators will evaluate the effect of stellate ganglion block on stress response of intubation in comparison to traditional antistress measures in adult patients

DETAILED DESCRIPTION:
Both groups will have the same general anesthesia procedure, patients in stellate block group will receive lidocaine in the stellate block will in control group patients will receive Na.Cl as placebo. primary outcome will be stress response to subsequent endotracheal intubation measure by changes in heart rate

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* General anesthesia with endotracheal intubation
* ASA I/II

Exclusion Criteria:

* Pregnancy
* Hypersensitivity to local anesthetics
* Coagulopathy
* Infection at site of injection
* Patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
heart rate | 5 minutes
  measured in beat/min.

SECONDARY OUTCOMES:
mean arterial blood pressure | 5 minutes
  measured in mm.Hg

CONTACTS AND LOCATIONS:
Overall Officials: abdelraheem Elawamy, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes